CLINICAL TRIAL: NCT02598401
Title: The British Osteonecrosis Study: A Prospective Multi-centre Study to Examine the Natural History of Osteonecrosis in Older Children, Teenagers and Young Adults With Acute Lymphoblastic Leukaemia and Lymphoblastic Lymphoma
Brief Title: The British Osteonecrosis Study
Acronym: BONES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Nadia laila Amin, Chief Investigator, University of Leeds
Other Study IDs: 185365
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Osteonecrosis
MeSH Terms: conditions — Osteonecrosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be obtained for future genetic analysis.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observation — Observational study with no intervention

SUMMARY:
The aim of this research is to examine the natural history of osteonecrosis in older children, teenagers and young adults with acute lymphoblastic leukaemia and lymphoblastic lymphoma within the UK. In addition to using and validating new, internationally agreed, standard definitions for osteonecrosis, this study will provide the data needed to develop a radiological classification which correlates with clinical status.

DETAILED DESCRIPTION:
Children, teenagers or young adults between the age of 10 (including the day of the 10th birthday) and 24 years 364 days (at the time of diagnosis) with a first diagnosis of acute lymphoblastic leukaemia or lymphoblastic lymphoma (T-NHL or SmIg negative precursor B-NHL) diagnosed under standard criteria are eligible for BONES.

The recruitment target is 50 over a 2 year period, which is based on an anticipated ascertainment target of 75%.

Information will be collected on basic demographics, presenting features and diagnosis at initial recruitment. Further data will be collected at the end of induction to ascertain treatment and response, along with results of relevant investigations performed in induction detailed below. Clinical information collected will include height, weight and puberty stage. At the four subsequent time points when MRI imagine is performed further data will also be collected, including a physiotherapy assessment using a structured assessment tool and child health assessment questionnaire, and biochemical information.

Investigations

The results of the following investigations, usually performed as part of the routine assessment, will be collected:

1. At diagnosis - highest white cell count, immunophenotype, cytogenetics, molecular results; albumin; lipid profile; vitamin D level, PTH, bone profile
2. At the end of induction - MRD result, flow cytometry from end of induction bone marrow; albumin; lipid profile plus results of additional investigations of vitamin D, PTH and bone profile if performed.

DEXA scans should be performed on all children >10y old and on treatment for ALL. It is recommended that a DEXA scan is performed at diagnosis and then annually. The results of these DEXA scans will be collected.

MRI of the hips, knees and ankles should comprise of unenhanced coronal T1 and STIR images as a minimum protocol. Knees and ankles can be imaged together. Where further information of a specific joint is needed pre-treatment additional sequences in different planes could be performed at the discretion of the participating centre. MRI will be performed at the following time points:

1. Within 4 weeks of diagnosis
2. At the end of delayed intensification
3. One year after the start of maintenance
4. Two years after the start of maintenance
5. Three years after the start of maintenance

In the event of the development of osteonecrosis the patient should be managed according to local protocols and at the discretion of their own consultant. Information on treatment will be collected.

Radiological review:

A central review panel consisting of Paediatric Radiologists with an interest in paediatric haematology will meet quarterly to review each MRI in order to agree the grade of osteonecrosis and noting specific features according to the study radiology proforma.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of acute lymphoblastic leukaemia or lymphoblastic lymphoma (T-NHL or SmIg negative precursor B-NHL)

Exclusion Criteria:

- inability to have MRI scans of lower limbs

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, teenagers or young adults between the age of 10 (including the day of the 10th birthday)and 24 years 364 days (at the time of diagnosis) with a first diagnosis of acute lymphoblastic leukaemia or lymphoblastic lymphoma (T-NHL or SmIg negative precursor B-NHL) diagnosed under standard criteria are eligible for BONES.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of osteonecrosis | 5 years
  The incidence of osteonecrosis in older children, teenagers and young adults being treated for acute lymphoblastic leukaemia (ALL) in the UK at different time points in their treatment.

SECONDARY OUTCOMES:
Risk factors for development of osteonecrosis. | 5 years
  The risk factors for progression and the development of symptomatic osteonecrosis in this population.
Radiological features for prediction of progression of osteonecrosis | 5 years
  specific radiological features that predict for either progression or regression in those with asymptomatic osteonecrosis

CONTACTS AND LOCATIONS:
Overall Officials: Nadia L Amin, MBChB, Principal Investigator — University of Leeds
Locations (4):
- United Kingdom (4):
  - Birmingham Children's Hospital, Birmingham
  - Leeds Children's Hospital, Leeds
  - St James's University Hospital, Leeds
  - Southampton Children's Hospital, Southampton

REFERENCES:
- [Derived] Amin N, Kinsey S, Feltbower R, Kraft J, Whitehead E, Velangi M, James B. British OsteoNEcrosis Study (BONES) protocol: a prospective cohort study to examine the natural history of osteonecrosis in older children, teenagers and young adults with acute lymphoblastic leukaemia and lymphoblastic lymphoma. BMJ Open. 2019 May 22;9(5):e027204. doi: 10.1136/bmjopen-2018-027204. PMID 31122988